CLINICAL TRIAL: NCT05110534
Title: Randomized Controlled Trial on an Supportive Caries Preventive Programme in Children Undergoing Dental General Anaesthesia
Brief Title: Supportive Caries Preventive Programme in Children Undergoing Dental General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Innovationsausschuss beim Gemeinsamen Bundesausschuss, (Innovationsfund) Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BB 078/17
Record Dates: First submitted 2021-11-03; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries in Children
Keywords: General anaesthesia; Children; Caries prevention; Pediatric dentistry

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator
Masking Description: The participants were randomly allocated to the test and control groups by a computer-generated random sequence prepared by a statistician, blinded to the recruiting person.The examiners were blinded regarding the group status of the children, as other practice personal had to perform the preventive sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Received two additional preventive oral hygiene appointments; one week before the general anaesthesia treatment and one week after the general anaesthesia.
  Interventions: Behavioral: additional oral hygiene appointments
- Control group (No Intervention): Received only standard prevention, without two additional preventive oral hygiene appointments before and after the general anaesthesia.

INTERVENTIONS:
Behavioral: additional oral hygiene appointments — Two additional preventive sessions including oral hygiene instructions one week before the date of the general anaesthesia treatment and at the control visit about a week after the general anaesthesia.
  Arms: Intervention group

SUMMARY:
Early childhood caries is a persistent problem often leading to dental treatment under general anaesthesia (GA). Thus, this study was to investigate the preventive effect of two additional intensive oral hygiene appointments before and after general anaesthesia.

In this randomized, controlled clinical trial, 408 children (age 2-5 years, mean 4.2+-1.04) intended for general anaesthesia were recruited and randomly assigned to the intervention and control groups with or without two additional intensive oral hygiene appointments before and after the general anaesthesia. At baseline and at 6-/12-month follow-ups, Approximal Plaque Index (API), gingiva Sulcus Bleeding Index (SBI), caries and initial caries index: initial, decayed, missing, filled, teeth (idmft) were recorded.

DETAILED DESCRIPTION:
Early Childhood Caries (ECC) is considered to be a global problem, as it is one of the most prevalent diseases in childhood. This leads to a severe problem in the caries risk children being highly affected by ECC, mostly also non-cooperative and from lower socio-economic background. The dental treatment for these pre-school children often requires general anaesthesia (GA), which is associated with health risks and considerable costs.

Thus, this study was to investigate the preventive effect of two additional intensive oral hygiene appointments before and after general anaesthesia.

After approval by the Ethics Committee at the University of Greifswald (No. BB 078/17), children with an age range from 2 to 5 years assigned for dental treatment under general anaesthesia were recruited.

After obtaining informed consent from the parents, the participants were randomly allocated to the test and control groups by a computer-generated random sequence prepared by a statistician, blinded to the recruiting person. Both groups received a baseline examination and the standard preventive program offered within the German National Health System consisting of explaining the etiology of caries and preventive approaches such as practical training of the parents in tooth brushing in their child as well as recommending fluoridated toothpaste and a reduction of cariogenic snacks. Finally fluoride varnish was applied. The test group received two additional preventive sessions including oral hygiene instructions using plaque disclosing agent, toothbrushing and fluoride application, one week before the date of the general anaesthesia treatment and at the control visit about a week after the general anaesthesia.

The baseline and follow-up examinations at 6 and 12 months recorded caries, fillings and missing teeth due to caries according to the World Health Organisation (WHO) criteria and it included initial caries lesions according to International Caries Detection and Assessment System (ICDAS 1-3). The subcomponents were also added up as initial, decayed, missing, filled, teeth/surfaces (idmft/idmfs). Due to the young age of the children, only primary teeth were of relevance.

In addition, the Approximal Plaque Index (API) and the gingiva Sulcus Bleeding Index (SBI) were taken. The examiners were blinded regarding the group status of the children, as other practice personal had to perform the preventive sessions.

Sample size calculation and statistical analyses:

The expected difference in new caries lesions between test and control groups was taken as an outcome parameter for sample size calculation. Previous regional studies had shown a mean caries development of 2 +-1.5 per year after the general anaesthesia. An intensive prevention program may result in a caries reduction of 30%, corresponding to 0.5-0.6 dmft less in the test group. With α being 0.05 and a power β of 0.80, 142 children were needed in each group, with a drop-out of 30% (62 children) this would mean a total sample size of 408 children at baseline.

The collected data were entered in Excel (Microsoft, USA), then transferred to Stata (Version 14.2; Stata Corp, College Station, USA) for further statistical analysis. Due to the large sample size and the randomization matching or data linkage analysis were not required, but a drop-out analysis was carried out to exclude a bias caused by attrition within the study. A modelling of continuous variables was carried out using restricted cubic splines. Mixed models were used for adjusting the analyses of changes within every group between baseline and recalls and between the two groups. Linear models were used for calculating the absolute effect and ordinal logistic regression for calculating the relative effect via odds ratios.

ELIGIBILITY:
Inclusion Criteria:

* 2-5 years old children attending dental treatment under general anaesthesia
* parental approval

Exclusion Criteria:

* children above 5 years old
* no parental approval

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 406 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Approximal Plaque Index (API) | 1 year
  an index to assess oral health by calculating the accumulated dental plaque on teeth surfaces
Gingiva Sulcus Bleeding Index (SBI) | 1 year
  an index to assess oral health by calculating the inflammation and bleeding of the gingiva sulcus
Caries and Initial Caries Index: decayed, missing, filled teeth (idmft) | 1 year
  WHO index to assess caries prevalence and caries status

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Alkilzy, PD Dr., Principal Investigator — Department of Preventive and Pediatric Dentistry, University of Greifswald; Christian Splieth, Prof. Dr., Study Chair — Department of Preventive and Pediatric Dentistry, University of Greifswald
Locations (1):
- Department of Preventive and Pediatric Dentistry, University of Greifswald, Greifswald, Germany